CLINICAL TRIAL: NCT04758780
Title: Prospective Phase II Pilot Study, Assessing Imaging Performance of 89Zirconium-labelled Girentuximab (89Zr-TLX250) PET-CT (Positron Emission Tomography/Computerized Tomography) in Metastatic Triple Negative Breast Cancer Patients
Brief Title: Imaging Performance Assessment of 89Zi-girentuximab (89Zr-TLX250) PET in Metastatic Triple Negative Breast Cancer
Acronym: OPALESCENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Telix Pharmaceutical (Unknown); SIRIC ILIAD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-2020-25
Record Dates: First submitted 2021-01-14; First posted 2021-02-17 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: carbonic anhydrase IX (CAIX); 89Zr- girentuximab; 89Zr-TLX250 PET/CT; Metastatic Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Monocentric, open prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-TLX250 PET/CT (Experimental): 89Zr-TLX250 PET/CT
  Interventions: Drug: 89Zr-TLX250

INTERVENTIONS:
Drug: 89Zr-TLX250 — 89Zr-TLX250 PET/CT
  Other Names: 89Zr-girentuximab

SUMMARY:
The purpose of this study is to evaluate the use of 89Zr-labeled girentuximab (89Zr-TLX250) as a novel, carbonic anhydrase IX (CAIX) targeted PET/CT tracer for the imaging of metastatic triple negative breast cancer (TNBC) patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of 89Zr-labeled girentuximab (89Zr-TLX250) as a novel, Carbonic Anhydrase IX (CAIX) targeted PET/CT tracer for the imaging of metastatic triple negative breast cancer (TNBC) patients.

TNBC patients are known to be rapidly progressive and have a poor prognosis. This poor prognosis is due to the lack of common breast cancer targets in TNBC. As TNBC expresses CAIX, this stuy will evaluate CAIX targeting by using a radiolabeled monoclonal antibody that recognizes carbonic anhydrase IX (CAIX) : 89Zr- girentuximab otherwise known as 89Zr-TLX250. Previous and ongoing studies have demonstrated the potential application of 89Zr-TLX250 as a new PET/CT imaging tracer for the detection of renal cancer.

After establishing the TNBC targeting properties of the 89Zr-TLX250 PET/CT imaging tracer, it should be interesting to develop a new targeted therapy using TLX250- radiolabeled with a therapeutic radionuclide such as 177Lutétium.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
* Female or male, Age ≥ 18 years at time of study entry.
* Primitive triple negative breast cancer proven histologically, defined according to the following criteria:

  * Estrogen receptors <10%.
  * And progesterone receptors <10%.
  * And Human Epidermal Growth factor Receptor 2 (HER2) not amplified or not overexpressed.
* Breast Cancer (BC) recurrence documented by conventional imaging and/or FDG PET/CT with at least one measurable metastatic lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) and/or PET Response Criteria In Solid Tumors (PERCIST).
* Consent to use a contraception method for at least 30 days after administration of 89Zr-TLX250.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Life expectancy at least 6 months.
* Patient has valid health insurance.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* History of another primary malignancy except for basal cell carcinoma within the last 5 years.
* Chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to the planned administration of 89Zr-TLX250 or continuing adverse effects (> grade 1) from such therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).
* Planned antineoplastic therapies (for the period between IV administration of 89Zr-TLX250 and imaging).
* Exposure to murine or chimeric antibodies within the last 5 years.
* Previous administration of any radionuclide within 10 half-lives of the same.
* Impossibility to hold lying motionless at least 1 hour, or known claustrophobia.
* Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune or metabolic), that may interfere with the objectives of the study or with the safety or compliance of the subject, as judged by the investigator.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Pregnant or likely to be pregnant or nursing patient.
* Known hypersensitivity to girentuximab or desferoxamine.
* Renal insufficiency with Glomerular Filtration Rate : GFR ≤ 45 mL/min/ 1.73 m².
* Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian.
* Disorder precluding understanding of trial information or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, Study Chair — Institut de Cancerologie de l'Ousest - ICO
Locations (1):
- ICO René Gauducheau, Saint-Herblain, France

REFERENCES:
- [Derived] Rousseau C, Heyman MF, Ferrer L, Rauscher A, Morel A, Rusu D, Frenel JS, Taupin M, Vilcot L, Allam N, Robert M, Campone M, Campion L, Kraeber-Bodere F. Prospective pilot study with [89Zr]Zr-girentuximab PET/CT: CA-IX imaging in metastatic triple negative breast cancer (OPALESCENCE). Eur J Nucl Med Mol Imaging. 2025 Nov 1. doi: 10.1007/s00259-025-07619-y. Online ahead of print. PMID 41174094

RESULTS

PARTICIPANT FLOW:
Groups:
- 89Zr-TLX250 PET/CT: Pretherapeutic 89Zr-TLX250 PET/CT
  89Zr-TLX250 PET/CT: Pretherapeutic 89Zr-TLX250 PET/CT
Period: Overall Study
Arm/Group | 89Zr-TLX250 PET/CT
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Metastatic triple negative breast cancer participants. Most patients received multiple treatments, with up to 4 treatments in combination (neoadjuvant and adjuvant chemotherapy, surgery and local radiotherapy).
  Of the 4 patients with immediate metastatic disease, 3 were enrolled without prior treatment, while the fourth received first-line targeted therapy.
Arm/Group | 89Zr-TLX250 PET/CT
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 68 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Total Lesions Detected on 89Zr-TLX250 PET/CT Versus 18FDG PET/CT
Description: The number of total lesions detected on 89Zr-TLX250 PET/CT versus 18FDG PET/CT is reported to assess the concordance for tumor lesion detection using 89Zr-TLX250 PET/CT and 18FDG) PET/CT
Time Frame: 5 days
Measure: Number; unit: lesions
Units Other Than Participants: all lesions
Groups:
- Number of Total Lesions Detected on 89Zr-TLX250 PET/CT Versus 18FDG PET/CT: The number of total lesions detected on 89Zr-TLX250 PET/CT versus 18FDG PET/CT is reported to assess the concordance for tumor lesion detection using 89Zr-TLX250 PET/CT and 18FDG) PET/CT
Arm/Group | Number of Total Lesions Detected on 89Zr-TLX250 PET/CT Versus 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (all lesions) | 273
lesions
  18FDG PET/CT | 264
  89Zr-TLX250 PET/CT | 231

2. Primary Outcome: Number of Brain Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of brain lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and 18FDG PET/CT.
  The detection performance of 89Zr-TLX250 PET/CT and 18FDG PET/CT for identifying brain lesions has been compared.
Time Frame: 5 days
Population: Only participants with brain lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT assessed for this Outcome Measure.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Brain Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of brain lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Brain Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 1
Number analyzed (lesions) | 3
lesions
  89Zr-TLX250 PET/CT | 3
  18FDG PET/CT | 1

3. Secondary Outcome: Tumor Burden Volume by 18FDG PET/CT and 89Zr-TLX250 PET/CT
Description: Total tumor burden (whole body) detected on 89Zr-TLX250 PET/CT scan compared to that defined on 18FDG PET/CT used as the reference performed at day 3 (D3) and at day 5 (D5)
Time Frame: 5 days
Measure: Median (Inter-Quartile Range); unit: cm3
Units Other Than Participants: lesions
Groups:
- Tumor Burden Volume by 18FDG PET/CT and 89Zr-TLX250 PET/CT: Total tumor burden (whole body) detected on 89Zr-TLX250 PET/CT scan compared to that defined on 18FDG PET/CT used as the reference performed at day 3 (D3) and at day 5 (D5)
Arm/Group | Tumor Burden Volume by 18FDG PET/CT and 89Zr-TLX250 PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 273
cm3
  89Zr-TLX250 PET/CT D3 | 41.01 [16.71 to 138.68]
  89Zr-TLX250 PET/CT D5 | 37.42 [24.70 to 173.75]
  18FDG PET/CT D3 | 41.21 [13.42 to 184.16]
  18FDG PET/CT D5 | 51.79 [29.17 to 103.26]

4. Secondary Outcome: Number of Patient With Concordance Between the 89Zr-TLX250 PET/CT Uptake and CAIX Histological Expression
Description: Number of patients with a concordance between the 89Zr-TLX250 PET/CT uptake and CAIX histological expression considered as positive or negative
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Number of Patients With Concordance Between the 89Zr-TLX250 PET and CAIX Histological Expression: Number of patients with a concordance between the 89Zr-TLX250 PET/CT uptake and CAIX histological expression considered as positive or negative
- Number of Patients With no Concordance Between the 89Zr-TLX250 PET and CAIX Histological Expression: Number of patients with no concordance between the 89Zr-TLX250 PET/CT uptake and CAIX histological expression considered as positive or negative
Arm/Group | Number of Patients With Concordance Between the 89Zr-TLX250 PET and CAIX Histological Expression | Number of Patients With no Concordance Between the 89Zr-TLX250 PET and CAIX Histological Expression
Number analyzed (Participants) | 12 | 12
Participants | 7 | 5

5. Secondary Outcome: Number of Participants With Adverse Events Related to 89Zr-TLX250
Description: All Adverse Events related to 89Zr-TLX250 are reported and assessed using CTCAE v5.0 scale
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Adverse Events Related to 89Zr-TLX250: All Adverse Events related to 89Zr-TLX250 are reported and assessed using CTCAE v5.0 scale
Arm/Group | Number of Participants With Adverse Events Related to 89Zr-TLX250
Number analyzed (Participants) | 12
Participants | 0

6. Secondary Outcome: Number of Participants With Serious Adverse Events Related or Not to 89Zr-TLX250
Description: All Serious Adverse Events are collected between the 89Zr-TLX250 administration and 30 days after. They assessed using CTCAE v5.0 scale
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Serious Adverse Events Related or Not to 89Zr-TLX250: All Serious Adverse Events are collected between the 89Zr-TLX250 administration and 30 days after. They assessed using CTCAE v5.0 scale
Arm/Group | Number of Participants With Serious Adverse Events Related or Not to 89Zr-TLX250
Number analyzed (Participants) | 12
Participants | 0

7. Primary Outcome: Number of Breast Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of breast lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Time Frame: 5 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Breast Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of breast lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Breast Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 25
lesions
  89Zr-TLX250 PET/CT | 25
  18FDG PET/CT | 23

8. Primary Outcome: Number of Bone Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of bone lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Time Frame: 5 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Bone Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of bone lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Bone Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 112
lesions
  89Zr-TLX250 PET/CT | 102
  18FDG PET/CT | 111

9. Primary Outcome: Number of Lymph Nodes Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of lymph nodes lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Time Frame: 5 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Lymph Nodes Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of lymph nodes lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Lymph Nodes Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 78
lesions
  89Zr-TLX250 PET/CT | 65
  18FDG PET/CT | 74

10. Primary Outcome: Number of Lung Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of lung lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Time Frame: 5 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Lung Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of lung lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Lung Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 27
lesions
  89Zr-TLX250 PET/CT | 17
  18FDG PET/CT | 27

11. Primary Outcome: Number of Liver Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Description: Number of liver lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Time Frame: 5 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Number of Liver Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT: Number of liver lesions seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT will be reported in order to evaluate the sensitivity of 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Arm/Group | Number of Liver Lesions Seen on 89Zr-TLX250 PET/CT and on 18FDG PET/CT
Number analyzed (Participants) | 12
Number analyzed (lesions) | 19
lesions
  89Zr-TLX250 PET/CT | 12
  18FDG PET/CT | 19

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated during 30 days after [89Zr]Zr-girentuximab administration
Description: All serious and non serious adverse events are collected
Arm/Group | 89Zr-TLX250 PET/CT
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04758780/Prot_SAP_000.pdf